CLINICAL TRIAL: NCT00547573
Title: A Multinational, Randomized, Double-Blind, Parallel, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tadalafil Administered "On Demand" to Asian Men With Erectile Dysfunction
Brief Title: Determine Safety and Effectiveness of Tadalafil in Asian Men When Taken as Needed for Getting and Keeping an Erection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5874; H6D-MC-LVDY
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): 10 mg tadalafil tablet
  Interventions: Drug: tadalafil
- 3 (Active Comparator): 20 mg tadalafil tablet
  Interventions: Drug: tadalafil
- 1 (Placebo Comparator): placebo tablet
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tadalafil — 10 mg tadalafil tablet taken by mouth as needed for 12 weeks not more than once a day
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: tadalafil — 20 mg tadalafil tablet taken by mouth as needed for 12 weeks not more than once a day
  Other Names: LY450190; Cialis; IC351
  Arms: 3
Drug: placebo — placebo tablet taken by mouth as needed for 12 weeks not more than once a day
  Arms: 1

SUMMARY:
Study to determine if tadalafil works better than placebo for Asian men having trouble getting or keeping an erection.

ELIGIBILITY:
Inclusion Criteria:

* History of erection problems
* Anticipate a monogamous female sexual relationship
* Abstain from other erection treatments at least 4 weeks before first dose and throughout the study
* Must be able to make required sexual intercourse attempts

Exclusion Criteria:

* Other primary sexual disorders
* History of radical prostatectomy or other pelvic surgery that affected being able to have an erection
* History of penile implant or clinically significant penile deformity
* Nitrate use
* Certain heart problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2003-04; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
IIEF Erectile Function Domain score from Questions 1-5 and 15. SEP Diary responses to Questions 2-3 and the entire Diary for baseline and endpoint scores. | 4, 8, and 12 weeks

SECONDARY OUTCOMES:
IIEF questions and scores, Global Assessment Questions, Patient's SEP Diary | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, ESt), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak to your personal physician., Beijing, China

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com